CLINICAL TRIAL: NCT00281203
Title: Innate and Adaptive Immunity in COPD Exacerbations: Bronchoscopies on Healthy Volunteers
Brief Title: Comparison of Alveolar Macrophages in Healthy Individuals Versus Individuals With COPD
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L. Curtis, Professor of Internal Medicine (Pulmonary & Critical Care Medicine), University of Michigan
Other Study IDs: 1327; R01HL082480 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy smokers: Must be free of serious diseases that might make it dangerous to undergo bronchoscopy.
  Interventions: Procedure: blood drawing; Procedure: fiberoptic bronchoscopy

INTERVENTIONS:
Procedure: blood drawing — blood will be drawn on the entry visit and will starting the intravenous (IV) line on the day of bronchoscopy
Procedure: fiberoptic bronchoscopy — A flexible instrument will be passed through the mouth and into the lungs. Portions of the lungs will be washed, by injecting and immediately suctioning out a small amount of fluid. The entire return will be used for research purposes, and no results will be reported to the participant. Bronchoscopy is performed once.

SUMMARY:
This study group forms the normal subject control group in an experiment designed to determine whether the alveolar macrophages (AMø) of patients with chronic obstructive pulmonary disease (COPD) show abnormal responsiveness to bacterial and viral products. Specifically, the study will determine the dose-response characteristics of AMø for production of interleukin (IL)-6, IL-18, and IL-23 (pro-inflammatory cytokines) on stimulation by purified lipopolysaccharide, a synthetic lipopeptide (PAM3-Cys), or poly I:C. These stimuli mimic the response to Gram-negative bacteria, Gram-positive bacteria, and RNA viruses, respectively. Results of the AMø from these healthy volunteers will be compared with AMø of COPD patients and smokers (or ex-smokers) with normal pulmonary function; those samples are being obtained during clinically indicated bronchoscopies under a separate consent form.

DETAILED DESCRIPTION:
BACKGROUND:

COPD is one of the most pressing healthcare problems facing our nation. Acute exacerbations of COPD (AE-COPD) are responsible for the bulk of healthcare costs, and much of the morbidity and decline in health status among individuals with this common disease. The lack of accepted animal models of AE-COPD necessitates novel approaches using human samples. Advances in the understanding of the pathogenesis have been slowed, in part, due to controversy as to how exacerbations should be defined. The prevailing paradigm has defined AE-COPD as event-based. Such definitions clearly identify groups of patients with accelerated loss of pulmonary function and increased mortality. However, limited data show that symptom-based definitions of AE-COPD also capture episodes inducing significant morbidity and functional decline, and hence of concern to patients. Fundamental mechanisms are lacking to explain AE-COPD defined by either means.

Controversy also surrounds triggers of AE-COPD. Bacteria and viruses are involved in some episodes, but the relative importance of each is intertwined with disputes over the definition of AE-COPD. Progress at linking specific pathogens to molecular pathogenesis has been slow, both due to their diversity, and to the high rates of bacterial colonization of patients with COPD, even in the stable state. Moreover, in many AE-COPD cases, no pathogen can be identified. Without negating the value of analyzing infections with specific species of pathogens, it appears that progress in molecular pathogenesis could be accelerated by focusing on unifying features of the pulmonary immune response during AE-COPD.

DESIGN NARRATIVE:

Bronchoscopies will be performed on healthy volunteers. Subjects are reimbursed $30 for the initial visit and $150 at completion of the bronchoscopy to help defray travel expenses and for the time spent participating as a volunteer.

ELIGIBILITY:
Inclusion criteria:

* Healthy individuals with normal pulmonary function as defined by AmericanThoracic Society criteria (entry spirometry)

Exclusion criteria:

* Unstable cardiovascular disease
* Other systemic disease in which survival of more than 2 years is unlikely
* Mental incompetence or active psychiatric illness
* Currently taking more than 20 mg/day of Prednisone
* Participation in another experimental protocol within 6 weeks of study entry
* Asthma
* Cystic fibrosis
* Clinically significant bronchiectasis
* Lung cancer
* Other inflammatory or fibrotic lung disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2005-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
alveolar macrophage functions in vitro | day of bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Curtis, Study Chair — University of Michigan at Ann Arbor
Locations (1):
- University of Michigan at Ann Arbor, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Freeman CM, Curtis JL, Chensue SW. CC chemokine receptor 5 and CXC chemokine receptor 6 expression by lung CD8+ cells correlates with chronic obstructive pulmonary disease severity. Am J Pathol. 2007 Sep;171(3):767-76. doi: 10.2353/ajpath.2007.061177. Epub 2007 Jul 19. PMID 17640964
- [Background] Freeman CM, Han MK, Martinez FJ, Murray S, Liu LX, Chensue SW, Polak TJ, Sonstein J, Todt JC, Ames TM, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Cytotoxic potential of lung CD8(+) T cells increases with chronic obstructive pulmonary disease severity and with in vitro stimulation by IL-18 or IL-15. J Immunol. 2010 Jun 1;184(11):6504-13. doi: 10.4049/jimmunol.1000006. Epub 2010 Apr 28. PMID 20427767
- [Background] Freeman CM, Martinez FJ, Han MK, Ames TM, Chensue SW, Todt JC, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Lung dendritic cell expression of maturation molecules increases with worsening chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1179-88. doi: 10.1164/rccm.200904-0552OC. Epub 2009 Sep 3. PMID 19729666
- [Background] Han MK, Agusti A, Calverley PM, Celli BR, Criner G, Curtis JL, Fabbri LM, Goldin JG, Jones PW, Macnee W, Make BJ, Rabe KF, Rennard SI, Sciurba FC, Silverman EK, Vestbo J, Washko GR, Wouters EF, Martinez FJ. Chronic obstructive pulmonary disease phenotypes: the future of COPD. Am J Respir Crit Care Med. 2010 Sep 1;182(5):598-604. doi: 10.1164/rccm.200912-1843CC. Epub 2010 Jun 3. PMID 20522794
- [Background] Curtis JL, Todt JC, Hu B, Osterholzer JJ, Freeman CM. Tyro3 receptor tyrosine kinases in the heterogeneity of apoptotic cell uptake. Front Biosci (Landmark Ed). 2009 Jan 1;14(7):2631-46. doi: 10.2741/3401. PMID 19273223
- [Background] Curtis JL, Freeman CM, Hogg JC. The immunopathogenesis of chronic obstructive pulmonary disease: insights from recent research. Proc Am Thorac Soc. 2007 Oct 1;4(7):512-21. doi: 10.1513/pats.200701-002FM. PMID 17878463
- [Result] Erb-Downward JR, Thompson DL, Han MK, Freeman CM, McCloskey L, Schmidt LA, Young VB, Toews GB, Curtis JL, Sundaram B, Martinez FJ, Huffnagle GB. Analysis of the lung microbiome in the "healthy" smoker and in COPD. PLoS One. 2011 Feb 22;6(2):e16384. doi: 10.1371/journal.pone.0016384. PMID 21364979
- [Result] Punturieri A, Copper P, Polak T, Christensen PJ, Curtis JL. Conserved nontypeable Haemophilus influenzae-derived TLR2-binding lipopeptides synergize with IFN-beta to increase cytokine production by resident murine and human alveolar macrophages. J Immunol. 2006 Jul 1;177(1):673-80. doi: 10.4049/jimmunol.177.1.673. PMID 16785566
- [Derived] Todt JC, Freeman CM, Brown JP, Sonstein J, Ames TM, McCubbrey AL, Martinez FJ, Chensue SW, Beck JM, Curtis JL. Smoking decreases the response of human lung macrophages to double-stranded RNA by reducing TLR3 expression. Respir Res. 2013 Mar 9;14(1):33. doi: 10.1186/1465-9921-14-33. PMID 23497334
- See also: COPD Foundation — http://www.copdfoundation.org/
- See also: Training Grant in Lung Diseases — http://www.med.umich.edu/intmed/pulmonary/edu/mtp.htm
- See also: Graduate Program in Immunology — http://www.med.umich.edu/immprog/